CLINICAL TRIAL: NCT02141425
Title: A Phase 1, Randomized, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP015K Following Single Doses in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP015K in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 015K-CL-HV07
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP015K
Keywords: Healthy volunteers; ASP015K
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP015K low dose (Experimental)
  Interventions: Drug: ASP015K
- ASP015K medium dose (Experimental)
  Interventions: Drug: ASP015K
- ASP015K high dose (Experimental): Optional, depending on safety review and regulatory authority input
  Interventions: Drug: ASP015K
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP015K — oral
  Arms: ASP015K high dose; ASP015K low dose; ASP015K medium dose
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single ascending doses of ASP015K.

DETAILED DESCRIPTION:
Subjects will be enrolled in 1 of 3 dose cohorts (low, medium and high). Each cohort will consist of 8 subjects with a 3:1 randomization ratio for ASP015K to placebo. Subjects will be confined to the clinic for study procedures until day 4 (5 days). After all subjects in a dose cohort have completed study procedures through day 4, a decision will be made whether or not dosing and enrollment of the next dose cohort should occur, which will only take place after a review of the safety and tolerability data through day 4 of the most recent dose cohort and any additional reported adverse events (AEs) for previously dosed cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be either:

  * Of non-childbearing potential:

    1. postmenopausal (defined as at least 1 year without any menses) prior to screening,
    2. or documented surgically sterile or status post-hysterectomy (at least 1 month prior to screening).
  * Or, if of childbearing potential:

    1. must have a negative pregnancy test at screening and day -1.
    2. must use highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and throughout the study period and for 90 days after final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 90 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the study period, and for 90 days after final study drug administration.
* Male subject must not donate sperm starting at screening and continuing throughout the study period, and for 90 days after final study drug administration.
* Subject has a Body Mass Index (BMI) range of 18.5 to 32.0 kg/m2, inclusive, and must weigh at least 50 kg at screening.
* Subject must be capable of swallowing multiple (up to 20) tablets.
* Subject agrees not to participate in another investigational study while on treatment.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months before screening assessment or breast feeding within 3 months before screening.
* Subject has a known or suspected hypersensitivity to ASP015K or any components of the formulations used.
* Subject has any of the liver function tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase or total bilirubin) above the ULN at screening or day -1. If the result is outside the limits, the assessment may be repeated once at screening and day -1.
* Subject has any clinically significant history of allergic conditions.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal (GI), endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy, as judged by the investigator or designee.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (non-cutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse < 40 or > 90 beats per minute, mean systolic blood pressure (BP) > 140 mmHg or mean diastolic BP > 90 mmHg (measurements taken in triplicate after subject has been resting in sitting position for 5 minutes) at screening or day -1.
* Subject has a mean QTcF interval of > 430 msec (for males) and > 450 msec (for females) at screening or day -1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken. If this triplicate also gives an abnormal result, the subject should be excluded.
* Subject has used any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, with the exception of hormone replacement therapy (HRT), hormonal contraceptives and intermittent acetaminophen (no more than 2g per day).
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past 6 months prior to screening.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical substance abuse within the past 2 years prior to screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* Subject has a positive test for alcohol, drugs of abuse or cotinine at screening or day -1.
* Subject anticipates an inability to abstain from xanthine (e.g., caffeine), grapefruit, Seville oranges (including marmalade), star fruit or any products containing these items from 72 hours prior to day -1 and throughout the duration of the study.
* Subject has used any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to day -1.
* Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive test for hepatitis B surface antigen, anti-hepatitis A virus (Immunoglobulin M) antibody, anti-hepatitis C virus antibody, hepatitis B core antibody or anti-human immunodeficiency virus Type 1 or Type 2 at screening.
* Subject has a positive tuberculosis skin test, Quantiferon Gold® or T-SPOT® test at screening.
* Subject has received any vaccine within 60 days prior to study drug administration.
* Subject has an absolute neutrophil count (ANC) < 2000 cells/mm3 or a creatine phosphokinase (CPK) > 1.5 x ULN at screening or day -1. If the result is outside the limits, the assessment may be repeated once at screening and day -1.
* Subject has had major GI surgery or has a medical condition that may inhibit the absorption and/or metabolism of study drug.
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives of the drug, whichever is longer, prior to screening.
* Subject has any other condition, which in the opinion of the investigator, precludes the subject's participation in the study.
* Subject is an employee of the Astellas Group, Janssen Pharmaceuticals or vendors involved in the study.
* Subject has participated in a prior study with ASP015K.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events, clinical laboratory tests, electrocardiogram (ECG) measurements, physical examination abnormalities and vital signs | Days 1-4

SECONDARY OUTCOMES:
Pharmacokinetic profile of ASP015K: Cmax, AUClast, AUCinf, tmax, t1/2, CL/F, Vz/F | Days 1-4
  Maximum Concentration (Cmax), Area Under the Plasma Concentration - Time Curve from Time Zero to Time of Last Measurable Concentration (AUClast), Area Under the Plasma concentration - Time Curve from Time Zero to Infinity (AUCinf), Time of Attain Cmax (tmax), Apparent Terminal Elimination Half-life (t1/2), Apparent total systemic clearance (CL/F), apparent volume of distribution (Vz/F)
Pharmacokinetic profile of ASP015K metabolites: Cmax, AUClast, AUCinf, tmax, t1/2 | Days 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- California Clinical Trials Medical Group/Parexel, Glendale, California, United States